CLINICAL TRIAL: NCT00810186
Title: Continuous Monitoring of Lungs Ventilation Dynamics by Small Surface Patches That Include Safe Mechanical Sensors. A Multicenter Study.
Brief Title: Continuous Monitoring of Lung Ventilation
Status: Completed | Type: Observational
Sponsor: Pneumedicare Ltd. (Industry)
Collaborators: Carmel Medical Center (Other); Bnai Zion Medical Center (Other Government); Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: NEO-01/2008
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Distress Syndrome, Newborn; Pulmonary Ventilation; Newborn, Abnormal; Apnea; Respiration Disorders
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Antisocial Personality Disorder; Apnea; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Newborns needing respiratory monitoring: Premature and term newborn infants (male/female)

SUMMARY:
Background: Patients that suffer from respiratory failure and need mechanical ventilation are at risk of further deterioration due to complications induced by progression of lung disease or the mechanical ventilation. The complications usually develop in a progressive manner, but are currently detected relatively late, when there is already severe and life threatening deterioration in patient oxygenation and sometimes irreversible damages.

Objective:To measure chest wall dynamics, derived from sensors placed on the chest and abdomen.

Methods: The system comprises of patches attached to the chest wall and upper abdomen that include mechanical sensors that measure the mechanics of lung inflation and deflation.

DETAILED DESCRIPTION:
Patients that suffer from respiratory failure and need mechanical ventilation are at risk of further life threatening deterioration following the development of mechanical problems related to airway management, development of lung barotrauma or displacement of the endotracheal tube.

Neonates especially need tight and sensitive monitoring of lung ventilation, because of the high prevalence of lung disease and need for ventilatory support in this population.

Methods:

The system comprises of patches attached to the chest wall and to the epigastrium. The patches include sensors that measure the mechanics of the lung inflation and deflation.

Study protocol

* Following parental informed consent, three patches will be placed on both sides of the chest and over the epigastric area in infants that require tight respiratory monitoring.
* The patches will be placed just beside the ECG patches.
* The placement of the patches will be performed by a physician.
* The monitoring can be preformed as long as the baby needs a tight respiratory monitoring. The patches will be replaced according to routine replacement policy of patches in the neonatal intensive care units, and at the regular time defined by the attending staff, and no longer than 24 hours. At the end of the data acquisition, the patches will be removed.
* No additional intervention is required.
* The patient will be inspected by the supervising physician involve in the research.
* It will not provide any data that may alter the treatment and will not interfere or influence the other monitoring devices that are used to evaluate the clinical status of the patient.
* The other parameters that are regularly monitored, that are displayed on the bedside monitor and respirator will be recorded by the research assistant. The ventilated baby will be identified by a study number. There will be a separate database for the measurements and the demographic and clinical data. There will be no disclosure of the patient's identity along with the data analysis and publication of the results or communication to authorities or other medical practitioners.

Equipment safety:

The system is safe for the use in human subjects. The whole system is approved for safety according to the acquired standard ICE-60601

ELIGIBILITY:
Inclusion Criteria:

* Infants that require tight monitoring of lung ventilation.
* Parents that understand and read Hebrew or Russian or Arabic.

Exclusion Criteria:

* Parental refusal to participate in the study.
* Premature babies under 700 grams.
* Prematurity below 26 weeks gestation.
* Severe edematous babies (Hydrops fetalis).
* Severe Hypoxic Ischemic Encephalopathy, initial brain injury or severe intracranial bleeding.
* Skin reactions to the adhesive patches.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants that require tight monitoring of lung ventilation admited to the Neonatal Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
A data-bank of the recordings obtained at various clinical settings acquired by the sensors | one year

SECONDARY OUTCOMES:
Establishment of a novel data bank that includes clinical cases of changes in ventilation and the comparison between the different monitored parameters. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dan Waisman, MD, Study Director — Department of Neonatology Carmel Medical Center
Locations (3):
- Israel (3):
  - Bnai Zion Medical Center, Haifa
  - Department of Neonatology, Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Haifa